CLINICAL TRIAL: NCT01437306
Title: A Single-Dose, Open-Label, Randomized, Two-Way Crossover Food Effect Study of Lofexidine 400 μg (2 x 200 μg) Tablets
Brief Title: Lofexidine Food Effect Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: USWM-LX1-1004; 1R01DA030916-01 (Other Grant/Funding Number: NIDA)
Record Dates: First submitted 2011-09-13; First posted 2011-09-20 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: lofexidine; food effect; pharmacokinetics; healthy volunteer
MeSH Terms: interventions — lofexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lofexidine following overnight fast (Experimental): A single dose of lofexidine (400 mcg or 2 x 200 mcg tablets) will be given to subjects following a minimum 10 hour overnight fast.
  Interventions: Drug: Lofexidine HCl
- Lofexidine Following a High Fat Meal (Experimental): A single dose of lofexidine 400 mcg (or 2 x 200 mcg tablets) will be administered to subjects following a standard high-fat meal.
  Interventions: Drug: Lofexidine HCl

INTERVENTIONS:
Drug: Lofexidine HCl — 400 mcg (2 x 200 mcg tablets) administered orally as a single dose

SUMMARY:
The objective of this single-dose, open-label, randomized, two-period, two-way crossover, food-effect study is to evaluate the effect of food on the rate of absorption and oral bioavailability of a test formulation of lofexidine 400 μg (2 x 200 μg tablet) manufactured by US WorldMeds, LLC.

DETAILED DESCRIPTION:
This is a single-dose, open-label, randomized, two-period, two-way crossover, food-effect study in which 12 healthy adult subjects will receive two separate single-dose administrations of lofexidine 400 μg (2 x 200 μg tablet). In one study period, subjects will be administered the study treatment following an overnight fast of at least 10 hours. In the other study period subjects will fast overnight for at least 10 hours, then begin consuming an FDA standard high-calorie, high-fat breakfast meal 30 minutes prior to administration of the study drug.

Subjects will be assigned numbers in an ascending order, based on successful completion of the screening process.

Subjects will receive each of the treatments listed below in randomized fashion during the two treatment periods:

Treatment A: Test Formulation Lofexidine 400 μg Dose = 2 x 200 μg tablet administered under fasted conditions US WorldMeds, LLC

Treatment B: Test Formulation Lofexidine 400 μg Dose = 2 x 200 μg tablet administered under fed conditions US WorldMeds, LLC

Each drug administration will be separated by a washout period of at least seven days. Each dose will be orally administered along with 240 mL (8 fl. oz.) of room temperature tap water. After dosing, no food will be allowed until 4 hours post-dose. Except for the 240 mL of room temperature tap water provided with the dose, no water may be consumed for 1 hour prior through 1 hour post dose. Meals will be the same and scheduled at approximately the same times relative to dose for each study period.

In order to prevent adverse events (AEs) of hypotension, all subjects will have intravenous (IV) access established at each check-in and will be administered normal saline (NS) at a continuous rate of 150 cc/hour until 1 hour prior to each dose administration. The IV catheter will remain in place for at least 12 hours postdose so that additional fluid can be administered if needed. If symptoms or clinically significant hypotension persist, IV fluid administration may continue for more than 12 hours, until it is no longer needed as determined by the Investigator.

Subjects who withdraw from the study may be replaced. During each study period, 6 mL blood samples will be obtained prior to each dosing and following each dose at selected times through 48 hours post-dose. A total of 28 pharmacokinetic blood samples will be collected from each subject, 14 samples in each study period. Plasma pharmacokinetic samples will be analyzed for lofexidine using a validated analytical method. Appropriate pharmacokinetic parameters will be calculated for each formulation using non-compartmental methods. In addition, blood will be drawn and urine will be collected for clinical laboratory testing at screening and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must satisfy the following criteria to be considered for study participation:

  * Subject must be a male or non-pregnant, non-breastfeeding female.
  * Subject must be between 18 and 50 years of age (inclusive).
  * Subject's Body Mass Index (BMI) must be between 18 and 30 kg/m2 (inclusive), and subject must weigh a minimum of 50 kg (110 lbs).
* Female subjects must agree to use one of the following forms of birth control from screening until 14 days after completion of the study:

  * Vasectomized partner (at least 6 months prior to dosing)
  * Post-menopausal (at least 2 years prior to dosing)
  * Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) at least 6 months prior to dosing
  * Double barrier (diaphragm with spermicide; condoms with spermicide)
  * IUD (intrauterine device)
  * Abstinence (must agree to use a double barrier method if they become sexually active during the study)
  * Implanted or intrauterine hormonal contraceptives in use for at least 6 consecutive months prior to study dosing and throughout the study duration
  * Oral, patch, and injected contraceptives or vaginal hormonal device (i.e. NuvaRing®) in use for at least 3 consecutive months prior to study dosing and throughout the study duration.
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to start of any study-specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of each confinement period.
* Subject is willing and able to consume the entire high-calorie, high-fat breakfast meal in the designated timeframe required during the assigned study period.
* Subject's vital signs must be within the following ranges to be included: Vital signs measured sitting after 3 minutes rest; heart rate: 40-90 bpm; systolic BP: 110-140 mmHg; diastolic BP: 60-90 mmHg. Out-of-range vital signs may be repeated once. Predose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified sub-investigator) prior to study drug administration. The Principal Investigator or designee will verify the eligibility of each subject with out-of-range vital signs and document approval prior to dosing.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history, electrocardiogram (ECG), or clinical laboratory results at screening.
* History of any syncopal episode or seizures.
* Presence of acute disease state (eg, nausea, vomiting, fever, diarrhea) within 7 days prior to scheduled dose administration.
* History or presence of allergic or adverse response to lofexidine or related drugs.
* Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial (randomized subjects only) within 30 days prior to the first dose of study medication.
* Has used any over-the-counter (OTC) medication, including nutritional supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication, except hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication.
* Subjects that have discontinued the use of implanted, intrauterine, or injected hormonal contraceptives must not have used any for 6 months prior to the first dose of study medication.
* Subjects that have discontinued the use of oral, patch, or vaginal hormonal contraceptives must not have used any for 1 month prior to the first dose of study medication.
* Has been treated with any known drugs that are moderate or strong inhibitors/inducers of CYP enzymes such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication and that in the Investigator's judgment may impact subject safety or the validity of the study results.
* Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
* Has any prior history of substance abuse or treatment (including alcohol) within the past 2 years.
* Is a female with a positive pregnancy test result.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).
* Has a positive test for Hepatitis B surface antigen, Hepatitis C antibody, or Human Immunodeficiency Virus (HIV) at screening or has been previously treated for Hepatitis B, Hepatitis C, or HIV infection.
* Has orthostatic hypotension at screening defined as a drop in systolic blood pressure ≥ 20 mmHg or a fall in diastolic blood pressure ≥ 10 mmHg following a 2 minute stand. Out-of-range vital signs may be repeated once. Predose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified sub-investigator) prior to study drug administration. The Principal Investigator or designee will verify the eligibility of each subject with out-of-range vital signs and document approval prior to dosing.
* Subjects with a QTcF greater than 450 msec (males) or greater than 470 msec (females), at screening obtained after 10 minutes rest in a supine position using the ECG machine algorithm.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Comparative Profile Pharmacokinetics TimeFrame 0.5, 1, 2, 3, 4, 5, 7, 10, 16, 24, 30, 36 and 48 hours post dose for Cmax, Tmax, Area Under the Curve, Elimination Rate Constant and Elimination Half Life | 48 Hours Following Each Dose
  Samples will be analyzed for lofexidine concentration and calculations will be performed for the following: Cmax and Tmax will be taken directly from the data.
  The elimination rate constant, will be calculated as the negative of the slope of the terminal log-linear segment of the plasma concentration time curve.
  Elimination half-life (T½) as follows: T½ = ln(2) / λZ
  Area under the curve will be calculated using the linear trapezoidal method and extrapolated to infinity using:
  AUCinf = AUClast + Clast/ λZ where Clast is the final concentration LOQ.

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Gorodetzky, MD, PhD, Principal Investigator — US WorldMeds; James A Longstreth, PhD, Principal Investigator — US WorldMeds
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States